CLINICAL TRIAL: NCT00029822
Title: Long-Term, Efficacy and Safety of Alfuzosin 10 MG OD on the Risk of Acute Urinary Retention and the Need for Surgery in Patients With BPH. A Two Year, Randomized, Multicenter, Double-Blind, Parallel Group, Placebo-Controlled Study.
Brief Title: Clinical Trial in Males With BPH (Enlarged Prostate)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC4485; SL770499
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Urinary Retention; Prostatic Hyperplasia; Benign Prostatic Hypertrophy
Keywords: Acute Urinary Retention; AUR; Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy; BPH; Enlarged Prostate
MeSH Terms: conditions — Urinary Retention; Prostatic Hyperplasia | interventions — alfuzosin

INTERVENTIONS:
Drug: Alfuzosin (SL770499)

SUMMARY:
A study to determine the effect on prevention of Acute Urinary Retention (inability to urinate) in males with an enlarged prostate, also known as BPH.

* Free study-related medical care provided.

ELIGIBILITY:
* Has been suffering for at least 6 months with any of the following symptoms:
* daytime or nighttime urinary frequency
* urgent feeling to urinate
* difficulty starting urinary stream
* interruption of urinary stream
* feeling of incomplete urination
* Has not had a previous episode of acute urinary retention
* Has not been diagnosed with prostate cancer
* Has not had previous prostate surgery
* Is not an insulin-dependent diabetic

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1522 (Actual)
Dates: Start 2001-05; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
occurrence of first episode of acute urinary retention (AUR)

SECONDARY OUTCOMES:
need for benign prostatic hyperplasia (BPH)-related surgery, international prostate symptoms score (IPSS)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (54):
- United States (35):
  - Medical Affiliated Research Center, Inc, Huntsville, Alabama
  - San Diego Urology Center, La Mesa, California
  - San Bernardino Urology Associates, San Bernardino, California
  - San Diego Urological Medical Group, San Diego, California
  - Pacific Clinical Research, Santa Monica, California
  - Urology Research Options, Aurora, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Renstar Medical Research, Plantation, Florida
  - Urology Associates, Marietta, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Urology of Indiana, LLC, Indianapolis, Indiana
  - Maryland Prostate Cancer, Baltimore, Maryland
  - Maryland Urology Association, Towson, Maryland
  - Newton Wellesley Urology, Newton, Massachusetts
  - Lakeside Urology, P.C., Saint Joseph, Michigan
  - Se Urology Network, Southaven, Mississippi
  - Weill Cornell Medical Center, New York, New York
  - Advanced Clinical Trials, Eugene, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Center for Urologic Care, West Reading, Pennsylvania
  - Matrix Research, Greenville, South Carolina
  - Ut Medical Group, Inc., Memphis, Tennessee
  - Murfreesboro Medical Center, Murfreesboro, Tennessee
  - nTouch Research Corporation, Dallas, Texas
  - Urology Consultants, P.A., San Antonio, Texas
  - Urology Associates, Fredericksburg, Virginia
  - Jeffrey Frankel, Seattle, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin
- Sanofi-aventis Administrative Office, Macquarie Park, Australia
- Sanofi-aventis Administrative Office, Sofia, Bulgaria
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Hørsholm, Denmark
- Sanofi-aventis Administrative Office, Helsinki, Finland
- Sanofi-aventis Administrative Office, Athens, Greece
- Sanofi-aventis Administrative Office, Budapest, Hungary
- Israel (4):
  - Edith Wolfson Hospital, Holon
  - Sapir Med. Center - Meir General Hospital, Kfar Saba
  - Rabin Medical Center-Golda Campus, Petah Tikvah
  - Sourasky Med. Center-Ichilov Hospital, Tel Aviv
- Sanofi-aventis Administrative Office, Gouda, Netherlands
- Sanofi-aventis Administrative Office, Lysaker, Norway
- Sanofi-aventis Administrative Office, Warsaw, Poland
- Sanofi-aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-aventis Administrative Office, Bucharest, Romania
- Sanofi-aventis Administrative Office, Midrand, South Africa
- Sanofi-aventis Administrative Office, Barcelona, Spain
- Sanofi-aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Result] Roehrborn CG. Alfuzosin 10 mg once daily prevents overall clinical progression of benign prostatic hyperplasia but not acute urinary retention: results of a 2-year placebo-controlled study. BJU Int. 2006 Apr;97(4):734-41. doi: 10.1111/j.1464-410X.2006.06110.x. PMID 16536764
- See also: Related Info — http://centerwatch.com
- See also: Related Info — http://www.sanofi-aventis.com